CLINICAL TRIAL: NCT01633463
Title: A Prospective Observational Study of Assessment of Pain and Its Treatment Adequacy in Emergency Department at Tertiary Care Cancer Hospital.
Brief Title: An Observational Study of Pain Assessment and Treatment Adequacy of Emergency Cancer Pain
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, DR. SWAPNIL YESHWANT PARAB, DR. SWAPNIL YESHWANT PARAB, Tata Memorial Hospital
Other Study IDs: emcap 2011
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: OBSERVE PAIN MANAGEMENT PRACTICES IN EMERGENCY DEPARTMENT
Keywords: EMERGENCY CANCER PAIN, ASSESSMENT, TREATMENT ADEQUACY.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
EMERGENCY CANCER PAIN DRAWS CANCER PATIENT TO EMERGENCY DEPARTMENT FOR TREATMENT. HOWEVER, THERE HAS BEEN INCONSISTENCY AND INADEQUACY OF PAIN MANAGEMENT IN EMERGENCY DEPARTMENT. THIS STUDY OBSERVES THE STATUS OF PAIN ASSESSMENT AND ITS ADEQUACY IN EMERGENCY DEPARTMENT IN A TERTIARY CARE CANCER HOSPITAL.

ELIGIBILITY:
Inclusion Criteria:

* ADULT CANCER PATIENTS REPORTING TO EMERGENCY DEPARTMENT WITH COMPLAINTS OF PAIN

Exclusion Criteria:

* 1.PATIENTS BELOW 18 YEARS OF AGE, 2. PATIENTS WITH INCOHERENT BEHAVIOUR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 ADULT CANCER PATIENTS REPORTING TO EMERGENCY DEPARTMENT WITH COMPLAINTS OF PAIN.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SWAPNIL Y PARAB, MD, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Hospital, Mumbai, Parel, Maharashtra, India